CLINICAL TRIAL: NCT01147146
Title: The Effects of Anesthetic Method on Cerebral Oxygen Saturation in Geriatric Patients Undergoing Transurethral Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Jeong-Yeon Hong / Associate Clinical Professor, Yonsei University, College of Medicine
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 4-2010-0133
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Surgery
Keywords: transurethral surgery
MeSH Terms: interventions — Propofol; Fentanyl; Atracurium; Bupivacaine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: propofol, fentanyl, atracurium — general anesthesia
  Other Names: propofol 2mg/kg, fentanyl 50mg, atracurium 0.5mg/kg
Drug: bupivacaine — spinal anesthesia
  Other Names: bupivacaine 8-10mg
Drug: bupivacaine, Midazolam — spinal anesthesia & sedation
  Other Names: Bupivacine 8-10mg, Midazolam 0.5mg/kg

SUMMARY:
The effects of anesthetic method on cerebral oxygen saturation in geriatric patients undergoing transurethral surgery.

ELIGIBILITY:
Inclusion Criteria:

* male patients (ASA physical status I and II) aged over 65 yrs and scheduled elective transurethral surgery

Exclusion Criteria:

* cardiovascular, renal, liver disease, or cerebrovascular disorder

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Yeon Hong, MD, Principal Investigator — Anesthesiology & Pain Medicine, Severance Hospital
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea